CLINICAL TRIAL: NCT04662411
Title: Butyrate/Hexanoate-enriched Triglycerides for Metabolic Health
Brief Title: Butyrate/Hexanoate in Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NL75253.068.20
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Metabolic Disease
MeSH Terms: conditions — Metabolic Diseases | interventions — Butyrates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- butyrate and hexanoate amount 1 (Experimental): 1325 mg of butyrate and hexanoate
  Interventions: Dietary Supplement: butyrate and hexanoate amount 1
- butyrate and hexanoate amount 2 (Experimental)
  Interventions: Dietary Supplement: butyrate and hexanoate amount 2
- butyrate and hexanoate amount 3 (Experimental)
  Interventions: Dietary Supplement: butyrate and hexanoate amount 3

INTERVENTIONS:
Dietary Supplement: Placebo — acute intake of 0 mg butyrate and hexanoate
  Arms: Placebo
Dietary Supplement: butyrate and hexanoate amount 1 — acute intake of 650 mg butyrate and hexanoate
  Arms: butyrate and hexanoate amount 1
Dietary Supplement: butyrate and hexanoate amount 2 — acute intake of 1325 mg butyrate and hexanoate
  Arms: butyrate and hexanoate amount 2
Dietary Supplement: butyrate and hexanoate amount 3 — acute intake of 2000 mg butyrate and hexanoate
  Arms: butyrate and hexanoate amount 3

SUMMARY:
In this study, we aim to identify a well consumable butyrate/hexanoate-enriched oil that increases circulating SCFA concentrations and improves postprandial substrate metabolism, which could be further used for a long-term study.

ELIGIBILITY:
Inclusion criteria

* Overweight/obese men (BMI ≥ 25 kg/m2 and ≤ 34.9 kg/m2);
* Aged 40 - 70 years;
* Caucasian;
* Normal blood pressure (systolic blood pressure 100-140mmHg, diastolic blood pressure 60-90 mmHg);
* Weight stable for at least 3 months (± 2 kg).

Exclusion criteria

* Type 2 diabetes mellitus (defined as fasting plasma glucose ≥ 7.1 mmol/L)
* Gastroenterological diseases or abdominal surgery (gallbladder removal and appendix removal are allowed)
* Cardiovascular diseases, cancer, liver or kidney malfunction, disease with a life expectancy shorter than 5 years;
* Lactose intolerance or other disorders that affect digestion (such as celiac disease)
* Abuse of products; alcohol and drugs, excessive nicotine use defined as >20 cigarettes per day; and excessive alcohol use defined as (> 15 units/week)
* Plans to lose weight or following of a hypocaloric diet in the following three months;
* Regular supplementation of pre- or probiotic products (for example Yakult, Activia), use of pre- or probiotics 3 months prior to the start of the study;
* Intensive exercise training more than three hours a week;
* Use of any medication that influences glucose or fat metabolism and inflammation (i.e. betablockers, corticosteroids, statins or NSAIDs);
* Regular use of laxation products in 3 months prior start of study or during study period;
* Use of antibiotics in the last three months (antibiotics use can alter substantially the gut microbiota composition).
* Follow a vegan diet or vegetarian diet.

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Plasma butyrate concentrations | Fasting and postprandial butyrate will be measured before and up to 6 hours after intake of the supplement
  Plasma butyrate concentrations

SECONDARY OUTCOMES:
Circulating Glucose | Fasting and postprandial glucose will be measured before and up to 6 hours after intake of the supplement
  Circulating Glucose assessed in plasma
Circulating Free Fatty Acids | Fasting and postprandial Free Fatty Acids will be measured before and up to 6 hours after intake of the supplement
  Circulating Free Fatty Acids assessed in plasma
Circulating Glycerol | Fasting and postprandial Glycerol will be measured before and up to 6 hours after intake of the supplement
  Circulating Glycerol assessed in plasma
Circulating Triglycerides (TG) | Fasting and postprandial TG will be measured before and up to 6 hours after intake of the supplement
  Circulating Triglycerides assessed in plasma
Circulating insulin | Fasting and postprandial insulin will be measured before and up to 6 hours after intake of the supplement
  Circulating . insulin will be assessed in plasma
Breath H2 | Fasting and postprandial breath H2 will be measured before and up to 6 hours after intake of the supplement
  Breath H2 using Gastrolyzer

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Deuren T, Smolders L, Hartog A, Bouwman FG, Holst JJ, Venema K, Blaak EE, Canfora EE. Butyrate and hexanoate-enriched triglycerides increase postprandrial systemic butyrate and hexanoate in men with overweight/obesity: A double-blind placebo-controlled randomized crossover trial. Front Nutr. 2023 Jan 4;9:1066950. doi: 10.3389/fnut.2022.1066950. eCollection 2022. PMID 36687671